CLINICAL TRIAL: NCT07274397
Title: Assessment of Early Post-operative Nuclear Imaging in Neurosurgery: a Safety and Feasibility Study in Patients Operated for Glioblastoma
Acronym: EARLYBRAINPET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beta Emitting Accurate Monitored Systems (Industry)
Collaborators: Assistance Publique - Hôpitaux de Paris, FRANCE (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Beams_EBP_25; 2025-A01745-44 (Other: ANSM)
Record Dates: First submitted 2025-09-16; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma; Brain Tumors; Brain Imaging
Keywords: Glioblastoma; brain tumors; PET-MRI; 18F-DOPA; Radiotracer; Diagnostic Imaging; Nuclear Medicine
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: The study follows a single-group, open-label, prospective design. All participants will receive the same diagnostic intervention: an early post-operative PET-MRI using 18F-DOPA and gadolinium-based contrast agent. The aim is to assess feasibility, safety, and imaging performance without a control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early post-operative PET-MRI group (Other): Participants in this arm will undergo early post-operative PET-MRI imaging within 48 hours after surgical resection of a suspected glioblastoma. The imaging procedure includes a brain MRI with gadolinium-based contrast and a PET scan using 18F-DOPA as the radiotracer. Patients will be monitored for potential adverse events related to the imaging agents and for radiation exposure. No therapeutic intervention will be administered. The purpose of this diagnostic intervention is to assess feasibility, safety, and imaging performance in detecting residual tumor tissue.
  Interventions: Diagnostic Test: Early post-operative brain PET-MRI with 18F-DOPA and Gadolinium

INTERVENTIONS:
Diagnostic Test: Early post-operative brain PET-MRI with 18F-DOPA and Gadolinium — This intervention consists of a combined brain PET-MRI imaging session performed within 48 hours after surgical resection of a suspected glioblastoma. The PET scan uses 18F-DOPA as the radiotracer, administered intravenously at a dose of 2 MBq/kg, with static brain acquisition starting immediately post-injection. The MRI includes standard sequences and gadolinium-based contrast-enhanced imaging. The goal is to assess the feasibility and safety of this early post-operative imaging procedure, and to validate imaging parameters for the detection of residual tumor. Radiation dosimetry and potential adverse events related to imaging agents will be monitored.

SUMMARY:
This clinical trial aims to evaluate the feasibility and safety of early post-operative brain PET-MRI imaging in adult patients who have undergone surgery for suspected glioblastoma. The study also seeks to validate specific nuclear imaging parameters for better detection of residual tumor tissue compared to standard gadolinium-enhanced MRI. The main objectives are to determine whether early PET-MRI within 48 hours post-surgery is feasible, to assess potential side effects related to imaging procedures, and to explore if PET parameters such as SUVmax, metabolic volume, and tumor-to-striatum ratio can improve the detection of tumor residue. A total of 15 patients will be included at a single site in France. Participants will undergo PET-MRI using 18F-DOPA and gadolinium, and will be monitored for radiation exposure and possible adverse events up to 24 hours after imaging.

DETAILED DESCRIPTION:
This study aims to assess safety and feasibility of early post-operative PET-MRI and validate imaging parameters for detecting glioblastoma residue, enabling future personalized post-surgical care.

The primary objectives are to :

* Asses the safety of performing early post-operative brain PET-MRI in neurosurgery patients after glioblastoma surgery.
* Measure the nuclear exposition of patients when performing early post-operative brain PET-MRI in neurosurgery patients.
* Assess the feasibility of performing early post-operative brain PET-MRI in neurosurgery patients.

It is a prospective interventional diagnostic study involving patient comparison Category RIPH. 15 patients will be included. This is a monocentric study. One surgical and including site (CHU Henri Mondor), in one country (France).

Patients will participate during 24 hours. The duration of the study is 12 months.

Following gadolinium injection, patients will be monitored for at least 30 minutes to allow for the early detection of potential side effects. Immediate hypersensitivity reactions, including anaphylactoid responses or other idiosyncratic effects, may present with cardiovascular, respiratory, or cutaneous symptoms, and can be severe.

Although delayed reactions are rare, most immediate events occur within the first 30 minutes post-administration. Monitoring is routinely implemented in clinical practice and will be applied accordingly in the study.

18F-DOPA injection can induce pain at the injection site, probably due to the acidity of the product. Given the minimal quantity of substance administered, the primary risk is associated with the exposure to ionizing radiation. In theory, such exposure may induce carcinogenesis or result in the development of hereditary defects. Nevertheless, since the effective dose is approximately 7 mSv and we are well below the maximum recommended activity of 280 MBq, the probability of these adverse effects occurring is considered very low.

2. MRI

1. Diffusion B1500
2. SWI
3. 3D FLAIR
4. 3D T1 SPACE
5. ASL
6. Spectroscopy (TE short et TE long) in the tumoral surroundings
7. After gadolinium injection : Perfusion T2*, Angio-MRI, 3DT1 SPACE

For PET-MRI imaging, tracer administration and acquisition timing will follow standard clinical protocols. For 18F-DOPA, a static brain acquisition will be performed between 10- and 30-minutes post-injection, as recommended for glioma imaging.

Study design is as follow :

• Pre-surgical baseline evaluation: 30 days - 2 days prior to surgery

* Patient information
* Medical History and Treatment, clinical assessment
* Preoperative Brain MRI and PET-MRI as detailed hereabove.

Patients usually undergo preoperative brain PET-MRI with gadolinium enhancement and 18F-DOPA injection as a standard of care. No specific period of time will be necessary to schedule the surgery after this imaging.

* D0: Neurosurgical procedure for tumor resection, as decided by the neurosurgeon, under general anesthesia
* Between D0 post-surgery and D2: patient informed consent and inclusion

  * H0: Patient informed consent and inclusion
  * Baseline medical examination
  * Patient transferred to the nuclear medicine department
  * Positioning of a dosimeter
  * Radiotracer intravenous injection
  * For suspected glioblastoma:

    18F-Dopa 2MBq/kg, starting the imaging immediately after injection
  * Postoperative brain PET-MRI acquisition
  * Surveillance time in nuclear medicine according to standard procedures
  * Patient transferred back to the neurosurgery department
  * Surveillance time: 24 hours dosimetry measurements
  * End of inclusion medical examination
  * Removing the dosimeter
  * H24: End of patient inclusion Neurosurgical follow-up and home discharge as established by the referent per clinical practice.

No medicinal product with therapeutic intent are administered in this study, only imaging agents usually used in clinical practice for diagnostic purposes are employed. The remainder of the patient's care will be managed according to the standard of care.

Only diagnostic imaging agents routinely used in standard clinical neuroimaging protocols will be administered during the study.

Gadolinium-based contrast agents will be used for MRI sequences requiring enhancement.

For PET imaging, 18F-DOPA will be employed. All imaging agents will be used under standard clinical conditions, in accordance with current safety and administration guidelines.

ELIGIBILITY:
Inclusion Criteria:

* First resection for a suspected glioblastoma in the past 72h
* Signed informed consent

non-inclusion Criteria:

* Deprived of liberty or under legal protection (e.g, guardianship, trusteeship)
* Patients under 18 years old
* Absence of social security cover
* Pregnancy
* Emergency procedure
* Contraindication to brain MRI, including claustrophobia
* Contraindication to radiotracers or gadolinium injection
* Preoperative cognitive impairment impeding patient information

Exclusion criteria :

* Any postoperative behavioral disorders or medical condition or symptom impeding the completion of brain imaging
* Postoperative medical dependency impeding the patient transfer to the nuclear medicine department (including, but not limited to, invasive ventilation, need for external ventricular drainage…)
* Postoperative histological diagnosis different from glioblastoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of performing early post-operative brain PET-MRI in neurosurgery patients | Within 24 hours after surgery
  by recording the rate of patients excluded after inclusion for non-realized imaging or incomplete imaging, at the physician's or the patient's demand.
Assess the safety of performing early post-operative brain PET-MRI in neurosurgery patients | Within 24 hours after surgery
  by collecting side effects associated with radiotracer injection and imaging procedure after surgery during the inclusion period
Assess the safety of performing early post-operative brain PET-MRI in neurosurgery patients | Whithin 24 hours after surgery
  by measuring ambient gamma dose rate at several time points (Hour 0, Hour 1, Hour 2, Hour 4 et Hour 24) on different points according to appendix.
Assess the safety of performing early post-operative brain PET-MRI in neurosurgery patients | Whithin 24 hours afin surgery
  by measuring ambient gamma dose rate at several time points on different points (on the patient, 50 centimeters, 1 meter, 2 meters from the patient) according to appendix.
Assess the safety of performing early post-operative brain PET-MRI in neurosurgery patients | Whithin 24 hours afin surgery
  With total dosimetry after 24 hours

SECONDARY OUTCOMES:
Validate a nuclear imaging protocol to measure residual tumor volume on early post-operative brain PET-MRI in neurosurgery patients | 24 hours
  by varying different parameters in PET analysis and comparing the results with gadolinium enhanced MRI: Dynamic analysis including peak time
Evaluate the inter-raters reliability of nuclear imaging protocol (T/S and T/CC) to evaluate the presence or absence of residual tumor on early post-operative brain PET in neurosurgery patients. | 24 hours
  Images will be reviewed by at least two raters : Kappa coefficient, Percentage agreement
Evaluate the inter-raters reliability of nuclear imaging protocol (metabolic volume with different thresholds) to measure residual tumor volume on early post-operative brain PET in neurosurgery patients. | 24 hours
  Intra-class correlation coefficient
Validate a nuclear imaging protocol to measure residual tumor volume on early post-operative brain PET-MRI in neurosurgery patients | 24 hours
  by varying different parameters in PET analysis and comparing the results with gadolinium enhanced MRI: Dynamic analysis including sleigh
Validate a nuclear imaging protocol to measure residual tumor volume on early post-operative brain PET-MRI in neurosurgery patients | 24 hours
  by varying different parameters in PET analysis and comparing the results with gadolinium enhanced MRI: Dynamic analysis including wash-out period
Validate a nuclear imaging protocol to measure residual tumor volume on early post-operative brain PET-MRI in neurosurgery patients | 24 hours
  by varying different parameters in PET analysis and comparing the results with gadolinium enhanced MRI: Standardized Uptake Value maximum
Validate a nuclear imaging protocol to measure residual tumor volume on early post-operative brain PET-MRI in neurosurgery patients | 24 hours
  by varying different parameters in PET analysis and comparing the results with gadolinium enhanced MRI: Tumour/Striatum ratio (T/S)
Validate a nuclear imaging protocol to measure residual tumor volume on early post-operative brain PET-MRI in neurosurgery patients | 24 hours
  by varying different parameters in PET analysis and comparing the results with gadolinium enhanced MRI: The rate of discordance between MRI result and PET result will be assessed for each modality